CLINICAL TRIAL: NCT06159010
Title: Relationship Between Renal Venous Return and Prognosis of Renal Function in Patients
Brief Title: Relationship Between Renal Venous Return and Prognosis of Renal Function in Patients With AKI in ICU
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICU-AKI
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Renal Venous Return
Keywords: Ultrasonography; Renal congestion; Renal venous flow; Intrarenal venous flow; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury
- Patients with non-acute kidney injury

SUMMARY:
A single-center prospective longitudinal observational study was carried out. Assessments were made on Days 1, 3, 5, and 7 after ICU admission in 90 patients with sepsis AKI, and 19 patients with septic without AKI only made assessments on Day 1. The primary outcome was CVP obtained at the time of renal ultrasonography. The association among RVF patterns, IRVF patterns, and CVP was examined using Student's t-test, and that with composite outcomes was assessed using a generalized estimating equation analysis, to account for intra-individual correlations.

DETAILED DESCRIPTION:
The prospective observational study was conducted at the ICU in China. The study was approved by the institutional review board of Peking Union Medical College Hospital (approval number, I-23PJ1176). All procedures were performed in accordance with the ethical standards of the local ethics committee on human experimentation and with the Helsinki Declaration of 1975.

Study participants

A single-center prospective longitudinal observational study is carried out at a tertiary critical care unit in China. Serial assessments were made of the renal RVF, IRVF, and CVP at 4-time points: Day one (D1) within 24 h of ICU admission, D1 + 48 h (D3), D1 + 96h (D5) and D1 + 144h (D7). Only adult patients (> 18 years) were included. AKI was staged using KDIGO criteria. Common to AKI research, the baseline creatinine value may not be known, and therefore defining AKI biochemically is not always possible. For those who had AKI defined using creatinine, we used the lowest value of any form within the 12 months prior to admission as a baseline value. If no preadmission creatinine was available, the lowest value the creatinine returned to after the resolution of acute illness was used. Failing all the above and if AKI could not be staged by other criteria, the admission creatinine was used as the baseline value. We excluded patients who (i) were on maintenance dialysis for chronic renal failure, (ii) were pregnant, (iii) had any ureteral obstructions because these affect the IRVF waveforms, and (vi) had earlier participation in this study.

Renal ultrasonography

The technical aspects of renal ultrasonography are as follows. Using a sector transducer, the right kidney in the left lateral supine position. Color Doppler images were used to determine a target renal and intrarenal vein. The RVF waveforms (the flow away from the transducer below the baseline) were classified into four waveform patterns: continuous or discontinuous (inclusion Biphasic continuous, Biphasic separated, and Monophasic). Specifically, a continuous pattern corresponded to the presence of continuous, uninterrupted venous flow below the baseline throughout the cardiac cycle, whereas the discontinuous pattern was a group of patterns that had at least one phase with zero velocity in venous flow during a cardiac cycle. The venous impedance index (VII), that is, the proportion of reduction in venous flow from its peak velocity (very low [0.2] in healthy subjects), was calculated as the peak maximum flow velocity minus the maximum flow velocity at the nadir in veins divided by the maximum flow velocity. The renal venous stasis index (RVSI) was calculated as the index cardiac cycle time minus the renal venous flow time divided by the index cardiac cycle time. In patients with sinus rhythm, we measured all indices over three cardiac cycles at the end of expiration and averaged them. In patients with atrial fibrillation, we measured the indices at a cardiac cycle where two preceding cardiac cycles had nearly equal durations. Echocardiography was performed at the bedside in the ICU. Meantime, CVP was measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients( > 18 years) were included. AKI was staged using KDIGO criteria. Common to AKI research, the baseline creatinine value may not be known and therefore defining AKI biochemically is not always possible. For those who had AKI defined using creatinine.

Exclusion Criteria:

* patients who were on maintenance dialysis for chronic renal failure, were pregnant, had any ureteral obstructions because these affect the IRVF waveforms, had earlier participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only adult patients (> 18 years) were included. AKI was staged using KDIGO criteria. Common to AKI research, the baseline creatinine value may not be known and therefore defining AKI biochemically is not always possible. For those who had AKI defined using creatinine, we used the lowest value of any form within the 12 months prior to admission as a baseline value. If no preadmission creatinine was available, the lowest value the creatinine returned to after the resolution of acute illness was used. Failing all the above and if AKI could not be staged by other criteria, the admission creatinine was used as the baseline value. We excluded patients who (i) were on maintenance dialysis for chronic renal failure, (ii) were pregnant, (iii) had any ureteral obstructions because these affect the IRVF waveforms, and (vi) had earlier participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
renal venous flow | Day 1,Day 3,Day 5, Day 7
intrarenal venous flow | Day 1,Day 3,Day 5, Day 7
center venous pressure | Day 1,Day 3,Day 5, Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, None Selected, China